CLINICAL TRIAL: NCT03185286
Title: 3D-Printed Personalized Metal Implant in Surgical Treatment of Ankle Bone Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Xiaojun Duan, Deputy Director of the Center for Joint Surgery, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3DIMPLANT
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Bone Diseases
Keywords: 3D printing, metal implant, bone defect
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D-printed personalized metal implant (Experimental): 3D-printed personalized metal implant will be used in bone defect surgeries.
  Interventions: Device: 3d-printed personalized metal implant

INTERVENTIONS:
Device: 3d-printed personalized metal implant — 3d-printed personalized metal implant will be used in subtalar arthrodesis.

SUMMARY:
This study aims to use 3D-printed personalized metal implants for bone defect surgeries in order to reduce pain of the patients.

DETAILED DESCRIPTION:
Bone defects are common in ankle disease, and the conventional treatment includes autologous or allogeneic bone grafts. However, autologous bone graft may cause complications and its source is rather limited; allogeneic bone graft may cause disease transmission and the mechanical strength of the graft is low after processing.

The 3D printing technology has provided a new way of solving this problem. It has the following technical advantages: wide range of graft sources, high mechanical strength, and can be prepared in advance according to various shapes.

Preparation procedure: first, establish the individualized ankle model according to the patient's ankle CT scan data and then prepare the implant model; second, conduct surgery rehearsal and place the implant model in the ankle model for observation; third, after confirmation, use titanium alloy in the 3D printing machine to prepare the individualized metal implant, which is in line with the Chinese National Standard "Wrought titanium and titanium alloy for surgical implants" (GB/T 13810-2007); fourth, implant the individualized metal implant into the bone defect area after sterilization.

ELIGIBILITY:
Inclusion Criteria:

* Receive ankle or subtalar arthrodesis;
* Refuse to use autologous bone graft or allogeneic bone graft.

Exclusion Criteria:

* The local defect area is small;
* Refuse to use permanent metal metal implant.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-12-31 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Postoperative 24 months
  The decrease in VAS score from baseline

SECONDARY OUTCOMES:
American Orthopedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Scale | Postoperative 24 months
  The increase in AOFAS score from baseline
Lower limb alignment | Postoperative 24 months
  Analyze the lower limb alignment by radiography
Osteotylus growth | Postoperative 24 months
  Analyze the osteotylus growth by radiography
Implant displacement | Postoperative 24 months
  Assess the implant displacement by radiography

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Duan, MD, Principal Investigator — Southwest Hospital, China
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No